CLINICAL TRIAL: NCT01478594
Title: A Phase 2, Open Label, Multicenter, Randomized Trial Comparing Tivozanib in Combination With mFOLFOX6 to Bevacizumab in Combination With mFOLFOX6, In Stage IV Metastatic Colorectal Cancer (mCRC) Subjects
Brief Title: A Study Combining mFOLFOX6 With Tivozanib or Bevacizumab in Patients With Metastatic Colorectal Cancer as First Line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4130-CL-0201; 2011-003502-24 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
Keywords: metastatic colorectal cancer; Avastin; bevacizumab; tivozanib; mFOLFOX6; BATON-CRC; AV951; ASP4130
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tivozanib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tivozanib + mFOLFOX6 (Experimental): Participants received 1.5 mg of tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received modified FOLFOX6 (mFOLFOX6) chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
  Interventions: Drug: Tivozanib; Drug: mFOLFOX6
- Bevacizumab + mFOLFOX6 (Active Comparator): Participants received a dose of 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
  Interventions: Drug: Bevacizumab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Tivozanib — Capsules for oral administration
  Other Names: AV951; ASP4130
  Arms: Tivozanib + mFOLFOX6
Drug: Bevacizumab — Solution for intravenous infusion
  Other Names: Avastin
  Arms: Bevacizumab + mFOLFOX6
Drug: mFOLFOX6 — mFOLFOX6 regimen is a combination therapy of oxaliplatin 85 mg/m^2 administered as an intravenous bolus over 2 hours on Days 1 and 15, leucovorin calcium 400 mg/m^2 administered as an intravenous bolus over 2 hours on Days 1 and 15, fluorouracil 400 mg/m^2 administered as an intravenous bolus over 5 to 15 minutes on Days 1 and 15, then 2400 mg/m^2 continuous intravenous infusion over 46 hours on Days 1 to 3 and 15 to 17.

SUMMARY:
The objective of this study is to compare the progression free survival (PFS), overall survival (OS), objective response rate (ORR), time to treatment failure (TTF), duration of response (DoR), quality of life, safety and tolerability of tivozanib in combination with mFOLFOX6 and bevacizumab in combination with mFOLFOX6.

DETAILED DESCRIPTION:
Imaging scans (computed tomography [CT]/magnetic resonance imaging [MRI]) to assess disease progression were to be completed within 28 days prior to first study drug administration, approximately every 8 weeks for the first 18 months and then approximately every 12 weeks until the patient showed progressive disease (PD) per the investigator, withdrew consent, was lost to follow-up or died. Per the original protocol, all patients were to be contacted by the study site every 12 weeks for survival following the end-of-treatment visit until death or for no more than 3 years after the end-of-treatment visit.

The interim futility analysis was conducted in December 2013, based on a pre-specified analysis cutoff date of 13 September 2013. The study was brought to a close as specified in the protocol due to the results of the interim futility analysis and only those participants who were deriving benefit (per the treating physician) from their current treatment remained on study until one of the discontinuation criteria was met.

Given the early closure of the study, no updated or additional efficacy analyses were performed after the interim analysis. A biomarker analysis was conducted in January 2014, based on the data from the cutoff date of 13 September 2013. The safety analysis was updated with a new cutoff date of 28 February 2014.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of metastatic colorectal cancer
* One measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* No prior systemic chemotherapy for advanced colorectal cancer; no fluorouracil containing adjuvant therapy in previous 6 months
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1

Exclusion Criteria:

* Any prior Vascular Endothelial Growth Factor (VEGF)-directed therapy or any other agent or investigational agent targeting the VEGF pathway
* Primary Central Nervous System (CNS) malignancies or CNS metastases
* Hematologic abnormalities:

  * Hemoglobin < 9.0 g/dL,
  * Absolute neutrophil count (ANC) < 2000 per mm^3,
  * Platelet count < 100,000 per mm^3,
  * Prothrombin (PT) or Partial Thromboplastin Time (PTT) > 1.5 X Upper Limit of Normal (ULN)
* Serum chemistry abnormalities:

  * Total bilirubin > 1.5 X ULN,
  * Aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT) > 2.5 X ULN,
  * Alkaline phosphatase > 2.5 X ULN,
  * Serum albumin < 2.0 g/dL,
  * Creatinine > 1.5 X ULN,
  * Proteinuria > 2+ by urine dipstick
* Significant cardiovascular disease
* Significant thromboembolic or vascular disorders within 6 months prior to administration of first dose of study drug
* Non-healing wound, bone fracture, or skin ulcer
* Inadequate recovery from any prior surgical procedure or major surgical procedure within 8 weeks prior to administration, or anticipation of major surgical procedure during the course of the study
* History of significant gastrointestinal (GI) toxicity, diarrhea, or stomatitis within the last 6 weeks
* An active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal condition with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug
* Serious/active infection or infection requiring antibiotics
* Significant bleeding disorders within 6 months prior to administration of first dose of study drug
* Active second primary malignancy, other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer and ductal or lobular carcinoma in situ of the breast. Subject is not considered to have a currently active malignancy if they have completed anti-cancer therapy and have been disease free for > 5 years
* History of allergic reactions, or intolerance, attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, history of Grade 3 hypersensitivity to oxaliplatin, history of allergic reaction to folic acid
* Female subject is pregnant or lactating
* Known history of genetic or acquired immune suppression disease including Human Immunodeficiency Virus (HIV); subjects on immune suppressive therapy for organ transplant
* Inability to swallow pills, malabsorption syndrome or gastrointestinal disease, major resection of the stomach or small bowel, or gastric bypass
* Uncontrolled neuro-psychiatric disorder or altered mental status
* Peripheral neuropathy ≥ Grade 2
* Participating in another interventional protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — AVEO Pharmaceuticals, Inc.
Locations (73):
- United States (27):
  - Banner MD Anderson Cancer Research Center, Gilbert, Arizona
  - Genesis Cancer Center, Hot Springs, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of California San Diego-Morris Cancer Center, La Jolla, California
  - UC Irvine Medical Center, Division of Hematology/Oncology, Orange, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - University of Florida, Davis Cancer Center (VA), Gainesville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Kaiser Foundation Hospitals, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Illinios Cancer Care, Peoria, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Associates of Oncology Hematology, P.C., Rockville, Maryland
  - University of Michigan Health, Ann Arbor, Michigan
  - NYU Cancer Institute, New York, New York
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Tri Country Hematology / Oncology, Canton, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Cancer Care Associates, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Oncology Hematology of Lehigh Valley, Bethlehem, Pennsylvania
  - Northern Utah Associates, Ogden, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (8):
  - St George Hospital, Kogarah, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ballarat Health Services, Ballarat, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Border Medical Oncology, Wodonga, Victoria
- Austria (3):
  - Medizinische Universitat Graz, Graz
  - Salzburger Landesklinken, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (4):
  - Ziekenhuisnetwerk Antwerpen - AZ Middelheim, Antwerp
  - Imelda VZW, Bonheiden
  - AZ Sint-Lucas Brugge, Bruges
  - AZ Groeninge - Campus Sint-Niklaas, Kortrijk
- Canada (5):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Hopital De La Cite-De-La-Sante, Laval, Quebec
  - Hopital Saint-Luc - Pavillon Principal, Montreal, Quebec
  - Chuq Centre Hospitalier Universitaire De Quebec, Québec, Quebec
- Czechia (2):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Finland (2):
  - Tampereen yliopistollinen sairaala, Tampere
  - Turun yliopistollinen keskussairaala, Turku
- Hungary (4):
  - Orszagos Onkologiai Intezet, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Gyula
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
- Italy (4):
  - Azienda Ospedaliero- Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Fondazione del Piemonte per I'Oncologia IRCC, Candiolo
  - IRCCS Azienda Ospedaliera Universitaria San Martino - Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Istituto Clinico Humanitas, Rozzano (MI)
- Amphia Ziekenhuis, Breda, Netherlands
- Spain (6):
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Corporacio Sanitaria Parc Tauli, Sabadell, Catalonia
  - Hospital Mutua de Terrassa, Terrassa, Catalonia
  - Centro Oncologico de Galicia, Galicia
  - Centro Integral Oncologico Clara Campal, Madrid
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Center, Glasgow
  - University College Hospital, London
  - Maidstone Hospital, Maidstone
  - Christie Hospital, Manchester
  - Peterborough and Stamford Hospitals NHS Foundation Trust, Peterborough

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were at least 18 years of age with Stage IV metastatic colorectal cancer (mCRC) and measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Version 1.1).
Pre-assignment Details: Participants were randomized in a 2:1 ratio (tivozanib to bevacizumab) and stratified by lactate dehydrogenase (LDH) status (< 1.5 x the upper limit of normal [ULN] or > 1.5 x ULN), origin of cancer (rectal or colon) and number of metastatic sites (1 or > 2).
Groups:
- Tivozanib + mFOLFOX6: Participants received 1.5 mg tivozanib orally once daily beginning on Day 1 of each 28-day cycle for 21 days followed by 7 days off treatment. Participants also received modified FOLFOX6 (mFOLFOX6) chemotherapy consisting of oxaliplatin, 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 bolus then 2400 mg/m^2 every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab + mFOLFOX6: Participants received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Period: Overall Study
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Started | 177 | 88
Treated | 177 | 87
Completed | 112 (Participants still on study as of 28 February 2014) | 60 (Participants still on study as of 28 February 2014)
Not Completed | 65 | 28
Not completed — Randomized but Never Received Study Drug | 0 | 1
Not completed — Death | 45 | 18
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Study Closed by Sponsor | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Tivozanib + mFOLFOX6: Participants received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Total: Total of all reporting groups
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6 | Total
Number analyzed (Participants) | 177 | 88 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.58) | 62.6 (11.17) | 62.2 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 33 | 92
  Male | 118 | 55 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 170 | 86 | 256
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 169 | 85 | 254
  Black or African American | 2 | 0 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or other Pacific Islander | 1 | 1 | 2
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 44 | 26 | 70
  Hungary | 24 | 8 | 32
  Czech Republic | 12 | 9 | 21
  Canada | 13 | 4 | 17
  Finland | 5 | 1 | 6
  Spain | 22 | 8 | 30
  Belgium | 10 | 9 | 19
  Austria | 8 | 3 | 11
  Australia | 15 | 9 | 24
  Netherlands | 1 | 1 | 2
  United Kingdom | 19 | 7 | 26
  Italy | 4 | 3 | 7
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG criteria: 0: Fully active. 1: Ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of all self-care. 3: Capable of limited self-care, confined to bed or chair more than 50% of waking hours. 4: Completely disabled, no self-care, totally confined to bed or chair. 5: Dead.
  participants
    ECOG Performance Status 0 | 95 | 58 | 153
    ECOG Performance Status 1 | 82 | 30 | 112
    ECOG Performance Status 2 | 0 | 0 | 0
    ECOG Performance Status 3 | 0 | 0 | 0
    ECOG Performance Status 4 | 0 | 0 | 0
Lactate dehydrogenase (LDH) Status [Number; unit: participants] — The upper limit of normal (ULN) from the site was used.
  participants
    < 1.5 Upper Limit of Normal | 127 | 64 | 191
    ≥ 1.5 Upper Limit of Normal | 50 | 24 | 74
Origin of Cancer [Number; unit: participants]
  Rectal | 53 | 24 | 77
  Colon | 124 | 64 | 188
Number of metastatic sites/organs [Number; unit: participants]
  1 | 56 | 30 | 86
  2 | 80 | 34 | 114
  3 | 29 | 21 | 50
  ≥ 4 | 12 | 3 | 15
Kirsten rat sarcoma (KRAS) Mutation Status [Number; unit: participants]
  Wild-type | 33 | 21 | 54
  Mutant | 23 | 16 | 39
  Unknown | 121 | 51 | 172
Time Since Initial Diagnosis [Mean (Standard Deviation); unit: months] | 9.41 (20.473) | 10.88 (21.055) | 9.90 (20.640)
Number of metastatic sites at screening [Mean (Standard Deviation); unit: metastatic sites] | 2.0 (1.02) | 2.0 (0.85) | 2.0 (0.97)

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Progression-Free Survival (PFS)
Description: The time from the date of randomization until objective tumor progression or death due to any cause. Objective tumor progression was determined through radiological imaging and based on the requirements of the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1):
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of existing non-target lesions or the appearance of one or more new lesions.
  Participants who did not progress or had not died at the time of the analysis were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: From randomization until the analysis cut-off date of 13 September 2013; median time on study drug was 167 days in the tivozanib group and 162 days in the bevacizumab group.
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6: Participants received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 177 | 88
months | 9.4 [8.5 to 10.1] | 10.7 [7.5 to 12.8]
Statistical Analysis 1: Comparison: Tivozanib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; An interim futility analysis was to be performed when approximately 83 PFS events (50% of the total PFS events) were observed. The Lans DeMets beta spending function with an O'Brien-Fleming boundary was used to derive the futility boundary. If the hazard ratio (HR) for PFS was greater than 1.0581, enrollment was to be stopped. With this futility stopping rule, the adjusted study power was 78.6%; Test type: Superiority or Other; p = 0.706, Log Rank; Stratification factors were LDH status (< 1.5 x ULN or ≥ 1.5 x ULN), origin of cancer (rectal or colon) and number of metastatic sites (1 or ≥ 2); Hazard Ratio (HR) = 1.091, 95% CI 2-sided [0.693 to 1.718] — HR presented for the stratified analysis, which was based on the Cox proportional hazards model. Assuming proportional hazards, an HR < 1 indicates a reduction in the HR in favor of tivozanib

2. Secondary Outcome: Progression-Free Survival (PFS) Based on Independent Radiological Review (IRR)
Description: The time from the date of randomization until the date of radiological disease progression assessed by the IRR or until death due to any cause, even in the absence of radiological progression.
Time Frame: 3 years
Population: Analysis was not performed due to study closure.
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the date of randomization until the documented date of death. Participants still alive at the time of analysis were censored on the last day the participant was known to be alive.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 177 | 88
months | NA [NA to NA] — Could not be estimated due to the low number of events at the time of the interim analysis | NA [12.8 to NA] — Could not be estimated due to the low number of events at the time of the interim analysis
Statistical Analysis 1: Comparison: Tivozanib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Test type: Superiority or Other; p = 0.754, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.116, 95% CI 2-sided [0.561 to 2.218] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) confirmed a minimum of four weeks apart based on RECIST 1.1 criteria.
  CR: Disappearance of all target and non-target lesions and no new lesions.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters and no progression of non-target lesions and no new lesions, or, disappearance of all target lesions and persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits and no new lesions.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number; unit: percentage of participants
Groups:
- Tivozanib + mFOLFOX6: Participants received 1.5 m tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 177 | 88
percentage of participants | 45.2 | 43.2
Statistical Analysis 1: Comparison: Tivozanib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Test type: Superiority or Other; p = 0.718, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) is defined as the time from the date of the first documented response of CR or PR (whichever is first recorded) to documented progression or death. If a participant did not progress or had not died at the time of analysis, the duration of response was censored at the date of last tumor assessment. Duration of response is only defined for participants whose best overall response was CR or PR.
Time Frame: as for outcome 1
Population: Participants with a best overall response of complete response (CR) or partial response (PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 80 | 38
months | 7.4 [5.6 to 11.3] | 9.3 [7.3 to 10.7]
Statistical Analysis 1: Comparison: Tivozanib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Test type: Superiority or Other; p = 0.437, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.389, 95% CI 2-sided [0.604 to 3.194] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to Treatment Failure (TTF) is defined as the time from randomization to last dose date of tivozanib/bevacizumab. If a participant discontinued treatment for any reason, the participant was considered as an event. Participants remaining on treatment at the time of analysis were censored at date of last dose.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 177 | 88
months | 5.5 [4.9 to 7.1] | 5.4 [3.7 to 6.7]
Statistical Analysis 1: Comparison: Tivozanib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Test type: Superiority or Other; p = 0.967, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.746 to 1.358] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Health Related Quality of Life (HRQoL)
Description: Time to deterioration in HRQoL measured by Colorectal cancer (CRC) subscale of the Functional Assessment of cancer Therapy Colorectal (FACT-C) scale, change in score from baseline using the European Quality of Life - 5 Dimensions (EQ-5D) and Fact Colorectal Symptom Index (FCSI) were not evaluated due to study closure.
Time Frame: 3 years
Population: Analysis was not performed due to study closure.
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Safety as Assessed by Physical Examination, Vital Signs, Laboratory Assessments, 12-lead Electrocardiogram (ECGs), and Adverse Events (AEs)
Description: An abnormality identified during a medical test is defined as an AE if the abnormality induced clinical signs or symptoms, required active intervention, interruption or discontinuation of study medication or was clinically significant in the investigator's opinion.
  An AE was serious if it resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly or birth defect, required or prolonged inpatient hospitalization or other medically important event.
  AEs, including abnormal clinical laboratory values, were graded using the National Cancer Institute Common Terminology Criteria for Grading Adverse Events (NCI-CTCAE) Version 4.03 per the following: 1=mild; 2= moderate; 3= severe; 4= life threatening; 5=death.
  Treatment-related AEs were defined as events where the relationship to study drug was marked as probably or possibly, or was missing.
Time Frame: From first dose through 30 days after last dose of either tivozanib or bevacizumab, until the data cut-off date of 28 February 2014. The median duration of treatment was 168.0 days in the tivozanib (tiv) arm and 162.0 days in the bevacizumab (bev) arm.
Population: The safety analysis set consisted of all randomized participants who received at least one dose of study drug (tivozanib or bevacizumab), analyzed according to the treatment actually received.
Measure: Number; unit: participants
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 177 | 87
participants
  Any adverse event | 177 | 87
  CTCAE Grade 3 or higher | 156 | 76
  Any tivozanib/bevacizumab-related adverse event | 158 | 74
  Any mFOLFOX6-related adverse event | 169 | 84
  Any tivozanib/bevacizumab and mFOLFOX6-related AE | 138 | 59
  Any tivozanib/bevacizumab-related AE ≥ Grade 3 | 104 | 31
  Any mFOLFOX6-related AE ≥ Grade 3 | 126 | 61
  Any tiv/bev and mFOLFOX6-related AE ≥ Grade 3 | 75 | 23
  Any AE with an outcome of death | 8 | 2
  Any tivozanib/bevacizumab-related AE of death | 3 | 2
  Any mFOLFOX6-related AE outcome of death | 3 | 2
  Any tiv/bev & mFOLFOX6-related AE outcome of death | 3 | 2
  Any serious adverse event (SAE) | 82 | 42
  Any tivozanib/bevacizumab-related SAE | 38 | 15
  Any mFOLFOX6-related SAE | 45 | 23
  Any tivozanib/bevacizumab and mFOLFOX6-related SAE | 30 | 11
  AE leading to tiv/bev discontinuation | 73 | 30
  AE leading to tivozanib/bevacizumab interruption | 138 | 63

9. Secondary Outcome: Progression-free Survival Events by Lactate Dehydrogenase (LDH) Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum lactate dehydrogenase status.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number; unit: participants
Groups:
- Tivozanib: LDH < 1.5 ULN: Participants with LDH status < 1.5 ULN received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: LDH ≥ 1.5 ULN: Participants with LDH status ≥ 1.5 ULN received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: LDH < 1.5 ULN: Participants with LDH status < 1.5 ULN received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab : LDH ≥ 1.5 ULN: Participants with LDH status ≥ 1.5 ULN received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: LDH < 1.5 ULN | Tivozanib: LDH ≥ 1.5 ULN | Bevacizumab: LDH < 1.5 ULN | Bevacizumab : LDH ≥ 1.5 ULN
Number analyzed (Participants) | 127 | 50 | 64 | 24
participants | 42 | 24 | 16 | 13
Statistical Analysis 1: Comparison: Tivozanib: LDH < 1.5 ULN vs Bevacizumab: LDH < 1.5 ULN; Test type: Superiority or Other; Hazard Ratio (HR) = 1.331, 95% CI 2-sided [0.746 to 2.375] — The hazard ratio was calculated using an unadjusted Cox proportional hazard model including treatment arms as the covariate. Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of Tivozanib arm
Statistical Analysis 2: Comparison: Tivozanib: LDH ≥ 1.5 ULN vs Bevacizumab : LDH ≥ 1.5 ULN; Test type: Superiority or Other; Hazard Ratio (HR) = 0.575, 95% CI 2-sided [0.285 to 1.160] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Progression-free Survival Events by Serum Vascular Endothelial Growth Factor-A (VEGF-A) Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum vascular endothelial growth factor-A (VEGF-A) level. VEGF-A protein levels were quantified using enzyme-liked immunosorbent assay (ELISA); the level of protein is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available serum protein samples
Measure: Number; unit: participants
Groups:
- Tivozanib: VEGF-A < Median: Participants with VEGF-A levels < median received 1.5 mg of tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: VEGF-A ≥ Median: Participants with VEGF-A levels ≥ median received 1.5 mg of tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-A < Median: Participants with VEGF-A levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-A ≥ Median: Participants with VEGF-A levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: VEGF-A < Median | Tivozanib: VEGF-A ≥ Median | Bevacizumab: VEGF-A < Median | Bevacizumab: VEGF-A ≥ Median
Number analyzed (Participants) | 54 | 54 | 29 | 26
participants | 20 | 24 | 6 | 12
Statistical Analysis 1: Comparison: Tivozanib: VEGF-A < Median vs Bevacizumab: VEGF-A < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.608, 95% CI 2-sided [0.635 to 4.073] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: VEGF-A ≥ Median vs Bevacizumab: VEGF-A ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.755, 95% CI 2-sided [0.375 to 1.521] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Progression-free Survival Events by Serum Vascular Endothelial Growth Factor-C (VEGF-C) Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum VEGF-C level. VEGF-C protein levels were quantified using enzyme-liked immunosorbent assay (ELISA); the level of protein is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available serum protein samples
Measure: Number; unit: participants
Groups:
- Tivozanib: VEGF-C < Median: Participants with VEGF-C levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: VEGF-C ≥ Median: Participants with VEGF-C levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-C < Median: Participants with VEGF-C levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-C ≥ Median: Participants with VEGF-C levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: VEGF-C < Median | Tivozanib: VEGF-C ≥ Median | Bevacizumab: VEGF-C < Median | Bevacizumab: VEGF-C ≥ Median
Number analyzed (Participants) | 52 | 56 | 27 | 28
participants | 15 | 29 | 8 | 10
Statistical Analysis 1: Comparison: Tivozanib: VEGF-C < Median vs Bevacizumab: VEGF-C < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.877, 95% CI 2-sided [0.366 to 2.100] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: VEGF-C ≥ Median vs Bevacizumab: VEGF-C ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.275, 95% CI 2-sided [0.614 to 2.646] — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Progression-free Survival Events by Serum VEGF-C / VEGF-A Ratio
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum VEGF-C/VEGF-A ratio. VEGF-A and VEGF-C protein levels were quantified using enzyme-liked immunosorbent assay (ELISA); the ratio is expressed relative to the observed median.
Time Frame: as for outcome 1
Population: Full analysis set with available serum protein samples
Measure: Number; unit: participants
Groups:
- Tivozanib: VEGF-C/VEGF-A < Median: Participants with VEGF-C/VEGF-A ratio < median received 1.5 mg of tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: VEGF-C/VEGF-A ≥ Median: Participants with VEGF-C/VEGF-A ratio ≥ median received 1.5 mg of tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-C/VEGF-A < Median: Participants with VEGF-C/VEGF-A ratio < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-C/VEGF-A ≥ Median: Participants with VEGF-C/VEGF-A ratio ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: VEGF-C/VEGF-A < Median | Tivozanib: VEGF-C/VEGF-A ≥ Median | Bevacizumab: VEGF-C/VEGF-A < Median | Bevacizumab: VEGF-C/VEGF-A ≥ Median
Number analyzed (Participants) | 53 | 55 | 26 | 29
participants | 21 | 23 | 11 | 7
Statistical Analysis 1: Comparison: Tivozanib: VEGF-C/VEGF-A < Median vs Bevacizumab: VEGF-C/VEGF-A < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.721, 95% CI 2-sided [0.345 to 1.507] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: VEGF-C/VEGF-A ≥ Median vs Bevacizumab: VEGF-C/VEGF-A ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.597, 95% CI 2-sided [0.672 to 3.795] — [estimate comment as in outcome 9, analysis 1]

13. Secondary Outcome: Progression-Free Survival Events by Soluble Vascular Endothelial Growth Factor Receptor-2 (sVEGFR-2) Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum sVEGFR-2 level. sVEGFR-2 protein levels were quantified using enzyme-liked immunosorbent assay (ELISA); the level of protein is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available serum protein samples
Measure: Number; unit: participants
Groups:
- Tivozanib: sVEGFR-2 < Median: Participants with sVEGFR-2 levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: sVEGFR-2 ≥ Median: Participants with sVEGFR-2 levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: sVEGFR-2 < Median: Participants with sVEGFR-2 levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: sVEGFR-2 ≥ Median: Participants with sVEGFR-2 levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: sVEGFR-2 < Median | Tivozanib: sVEGFR-2 ≥ Median | Bevacizumab: sVEGFR-2 < Median | Bevacizumab: sVEGFR-2 ≥ Median
Number analyzed (Participants) | 46 | 62 | 27 | 28
participants | 15 | 29 | 5 | 13
Statistical Analysis 1: Comparison: Tivozanib: sVEGFR-2 < Median vs Bevacizumab: sVEGFR-2 < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.627, 95% CI 2-sided [0.580 to 4.564] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: sVEGFR-2 ≥ Median vs Bevacizumab: sVEGFR-2 ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.779, 95% CI 2-sided [0.397 to 1.531] — [estimate comment as in outcome 9, analysis 1]

14. Secondary Outcome: Progression-Free Survival Events by Soluble Vascular Endothelial Growth Factor Receptor-3 (sVEGFR-3) Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum sVEGFR-3 level. sVEGFR-3 protein levels were quantified using enzyme-liked immunosorbent assay (ELISA); the level of protein is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available serum protein samples
Measure: Number; unit: participants
Groups:
- Tivozanib: sVEGFR-3 < Median: Participants with sVEGFR-3 levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: sVEGFR-3 ≥ Median: Participants with sVEGFR-3 levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: sVEGFR-3 < Median: Participants with sVEGFR-3 levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: sVEGFR-3 ≥ Median: Participants with sVEGFR-3 levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: sVEGFR-3 < Median | Tivozanib: sVEGFR-3 ≥ Median | Bevacizumab: sVEGFR-3 < Median | Bevacizumab: sVEGFR-3 ≥ Median
Number analyzed (Participants) | 50 | 58 | 30 | 25
participants | 14 | 30 | 4 | 14
Statistical Analysis 1: Comparison: Tivozanib: sVEGFR-3 < Median vs Bevacizumab: sVEGFR-3 < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.946, 95% CI 2-sided [0.636 to 5.956] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: sVEGFR-3 ≥ Median vs Bevacizumab: sVEGFR-3 ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.806, 95% CI 2-sided [0.422 to 1.538] — [estimate comment as in outcome 9, analysis 1]

15. Secondary Outcome: Progression-Free Survival Events by Serum Interleukin-8 (IL-8) Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum interleukin-8 level. IL-8 protein levels were quantified using enzyme-liked immunosorbent assay (ELISA); the level of protein is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available serum protein samples
Measure: Number; unit: participants
Groups:
- Tivozanib: IL-8 < Median: Participants with IL-8 levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: IL-8 ≥ Median: Participants with IL-8 levels ≥ median received 1.5 m tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: IL-8 < Median: Participants with IL-8 levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: IL-8 ≥ Median: Participants with IL-8 levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: IL-8 < Median | Tivozanib: IL-8 ≥ Median | Bevacizumab: IL-8 < Median | Bevacizumab: IL-8 ≥ Median
Number analyzed (Participants) | 53 | 55 | 27 | 28
participants | 14 | 30 | 7 | 11
Statistical Analysis 1: Comparison: Tivozanib: IL-8 < Median vs Bevacizumab: IL-8 < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.776, 95% CI 2-sided [0.303 to 1.991] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: IL-8 ≥ Median vs Bevacizumab: IL-8 ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.241, 95% CI 2-sided [0.615 to 2.501] — [estimate comment as in outcome 9, analysis 1]

16. Secondary Outcome: Progression-Free Survival Events by Serum Neuropilin Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline serum neuropilin level. Neuropilin protein levels were quantified using enzyme-liked immunosorbent assay (ELISA); the level of protein is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available serum protein samples
Measure: Number; unit: participants
Groups:
- Tivozanib: Neuropilin < Median: Participants with neuropilin levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: Neuropilin ≥ Median: Participants with neuropilin levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: Neuropilin < Median: Participants with neuropilin levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and FOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: Neuropilin ≥ Median: Participants with neuropilin levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: Neuropilin < Median | Tivozanib: Neuropilin ≥ Median | Bevacizumab: Neuropilin < Median | Bevacizumab: Neuropilin ≥ Median
Number analyzed (Participants) | 53 | 55 | 30 | 25
participants | 10 | 34 | 6 | 12
Statistical Analysis 1: Comparison: Tivozanib: Neuropilin < Median vs Bevacizumab: Neuropilin < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.950, 95% CI 2-sided [0.343 to 2.630] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: Neuropilin ≥ Median vs Bevacizumab: Neuropilin ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.983, 95% CI 2-sided [0.503 to 1.918] — [estimate comment as in outcome 9, analysis 1]

17. Secondary Outcome: Progression-Free Survival Events by Tumor VEGF-A Ribonucleic Acid (RNA) Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline tumor VEGF-A RNA level.
  RNA was purified from biopsy tissue and measured using quantitative reverse transcription polymerase chain reaction (qRT-PCR). Since low cycle threshold (CT) values reflect high RNA expression, the inverse of CT values were used to derive tumor categories. RNA level is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available tumor biopsy RNA samples
Measure: Number; unit: participants
Groups:
- Tivozanib: VEGF-A RNA < Median: Participants with VEGF-A RNA levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: VEGF-A RNA ≥ Median: Participants with VEGF-A RNA levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-A RNA < Median: Participants with VEGF-A RNA levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-A RNA ≥ Median: Participants with VEGF-A RNA levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: VEGF-A RNA < Median | Tivozanib: VEGF-A RNA ≥ Median | Bevacizumab: VEGF-A RNA < Median | Bevacizumab: VEGF-A RNA ≥ Median
Number analyzed (Participants) | 40 | 38 | 18 | 17
participants | 13 | 18 | 7 | 5
Statistical Analysis 1: Comparison: Tivozanib: VEGF-A RNA < Median vs Bevacizumab: VEGF-A RNA < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.226, 95% CI 2-sided [0.468 to 3.214] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: VEGF-A RNA ≥ Median vs Bevacizumab: VEGF-A RNA ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.232, 95% CI 2-sided [0.447 to 3.396] — [estimate comment as in outcome 9, analysis 1]

18. Secondary Outcome: Progression-Free Survival Events by Tumor VEGF-C RNA Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline tumor VEGF-C RNA level.
  RNA was purified from biopsy tissue and measured using quantitative reverse transcription polymerase chain reaction (qRT-PCR). Since low cycle threshold (CT) values reflect high RNA expression, the inverse of CT values were used to derive tumor categories. RNA level is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available tumor biopsy RNA samples
Measure: Number; unit: participants
Groups:
- Tivozanib: VEGF-C RNA < Median: Participants with VEGF-C RNA levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: VEGF-C RNA ≥ Median: Participants with VEGF-C RNA levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-C RNA < Median: Participants with VEGF-C RNA levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-A RNA ≥ Median: Participants with VEGF-C RNA levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: VEGF-C RNA < Median | Tivozanib: VEGF-C RNA ≥ Median | Bevacizumab: VEGF-C RNA < Median | Bevacizumab: VEGF-A RNA ≥ Median
Number analyzed (Participants) | 41 | 37 | 16 | 19
participants | 14 | 17 | 6 | 6
Statistical Analysis 1: Comparison: Tivozanib: VEGF-C RNA < Median vs Bevacizumab: VEGF-C RNA < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.803, 95% CI 2-sided [0.307 to 2.100] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: VEGF-C RNA ≥ Median vs Bevacizumab: VEGF-A RNA ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.505, 95% CI 2-sided [0.585 to 3.873] — [estimate comment as in outcome 9, analysis 1]

19. Secondary Outcome: Progression-Free Survival Events by Tumor VEGF-C / VEGF-A RNA Ratio
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline tumor VEGF-C/VEGF-A RNA ratio.
  RNA was purified from biopsy tissue and measured using quantitative reverse transcription polymerase chain reaction (qRT-PCR). Since low cycle threshold (CT) values reflect high RNA expression, the inverse of CT values were used to derive tumor categories. RNA level is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available tumor biopsy RNA samples
Measure: Number; unit: participants
Groups:
- Tivozanib: VEGF-C/VEGF-A RNA < Median: Participants with VEGF-C/VEGF-A RNA ratio < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: VEGF-C/VEGF-A RNA ≥ Median: Participants with VEGF-C/VEGF-A RNA ratio ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-C/VEGF-A RNA < Median: Participants with VEGF-C/VEGF-A RNA ratio < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-C/VEGF-A RNA ≥ Median: Participants with VEGF-C/VEGF-A RNA ratio ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: VEGF-C/VEGF-A RNA < Median | Tivozanib: VEGF-C/VEGF-A RNA ≥ Median | Bevacizumab: VEGF-C/VEGF-A RNA < Median | Bevacizumab: VEGF-C/VEGF-A RNA ≥ Median
Number analyzed (Participants) | 38 | 40 | 16 | 19
participants | 16 | 15 | 6 | 6
Statistical Analysis 1: Comparison: Tivozanib: VEGF-C/VEGF-A RNA < Median vs Bevacizumab: VEGF-C/VEGF-A RNA < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.356 to 2.385] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: VEGF-C/VEGF-A RNA ≥ Median vs Bevacizumab: VEGF-C/VEGF-A RNA ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.220, 95% CI 2-sided [0.462 to 3.220] — [estimate comment as in outcome 9, analysis 1]

20. Secondary Outcome: Progression-Free Survival Events by Tumor VEGF-D RNA Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline tumor VEGF-D RNA level.
  RNA was purified from biopsy tissue and measured using quantitative reverse transcription polymerase chain reaction (qRT-PCR). Since low cycle threshold (CT) values reflect high RNA expression, the inverse of CT values were used to derive tumor categories. RNA level is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available tumor biopsy RNA samples
Measure: Number; unit: participants
Groups:
- Tivozanib: VEGF-D RNA < Median: Participants with VEGF-D RNA levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: VEGF-D RNA ≥ Median: Participants with VEGF-D RNA levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-D RNA < Median: Participants with VEGF-D RNA levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: VEGF-D RNA ≥ Median: Participants with VEGF-D RNA levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: VEGF-D RNA < Median | Tivozanib: VEGF-D RNA ≥ Median | Bevacizumab: VEGF-D RNA < Median | Bevacizumab: VEGF-D RNA ≥ Median
Number analyzed (Participants) | 42 | 36 | 14 | 21
participants | 16 | 15 | 5 | 7
Statistical Analysis 1: Comparison: Tivozanib: VEGF-D RNA < Median vs Bevacizumab: VEGF-D RNA < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.915, 95% CI 2-sided [0.334 to 2.512] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: VEGF-D RNA ≥ Median vs Bevacizumab: VEGF-D RNA ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.384, 95% CI 2-sided [0.554 to 3.455] — [estimate comment as in outcome 9, analysis 1]

21. Secondary Outcome: Progression-Free Survival Events by Tumor Placental Growth Factor (PIGF) RNA Level
Description: The number of participants with a progression-free survival event (radiological progression assessed by the investigator or death due to any cause) reported by Baseline tumor PIGF RNA level.
  RNA was purified from biopsy tissue and measured using quantitative reverse transcription polymerase chain reaction (qRT-PCR). Since low cycle threshold (CT) values reflect high RNA expression, the inverse of CT values were used to derive tumor categories. RNA level is expressed relative to the observed median level.
Time Frame: as for outcome 1
Population: Full analysis set with available tumor biopsy RNA samples
Measure: Number; unit: participants
Groups:
- Tivozanib: PIGF RNA < Median: Participants with PIGF RNA levels < median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Tivozanib: PIGF RNA ≥ Median: Participants with PIGF RNA levels ≥ median received 1.5 mg tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: PIGF RNA < Median: Participants with PIGF RNA levels < median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
- Bevacizumab: PIGF RNA ≥ Median: Participants with PIGF RNA levels ≥ median received 5 mg/kg bevacizumab via intravenous infusion every 2 weeks on Days 1 and 15 of each cycle and mFOLFOX6 chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib: PIGF RNA < Median | Tivozanib: PIGF RNA ≥ Median | Bevacizumab: PIGF RNA < Median | Bevacizumab: PIGF RNA ≥ Median
Number analyzed (Participants) | 39 | 39 | 17 | 18
participants | 14 | 17 | 5 | 7
Statistical Analysis 1: Comparison: Tivozanib: PIGF RNA < Median vs Bevacizumab: PIGF RNA < Median; Test type: Superiority or Other; Hazard Ratio (HR) = 1.538, 95% CI 2-sided [0.548 to 4.320] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tivozanib: PIGF RNA ≥ Median vs Bevacizumab: PIGF RNA ≥ Median; Test type: Superiority or Other; Hazard Ratio (HR) = 0.744, 95% CI 2-sided [0.299 to 1.850] — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after last dose of either tivozanib or bevacizumab, until the data cut-off date of 28 February 2014. The median duration of treatment was 168.0 days in the tivozanib arm and 162.0 days in the bevacizumab arm.
Groups:
- Tivozanib + mFOLFOX6: Participants received 1.5 mg of tivozanib orally once daily beginning on Day 1 of each cycle for 21 days followed by 7 days off treatment. Participants also received mFOLFOX6) chemotherapy every 2 weeks on Days 1 and 15 of each cycle.
Arm/Group | Tivozanib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Serious Adverse Events (participants affected / at risk) | 82/177 | 42/87
Other Adverse Events (participants affected / at risk) | 175/177 | 85/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib + mFOLFOX6 (N=177) | Bevacizumab + mFOLFOX6 (N=87)
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 5 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 4 | 4
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Device related infection (Infections and infestations) | 2 | 3
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Perihepatic abscess (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 4 | 7
Disease progression (General disorders) | 3 | 0
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 1
Catheter site erythema (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Localised oedema (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Stent malfunction (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
Thrombosis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Amnesia (Nervous system disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Anorectal operation (Surgical and medical procedures) | 1 | 0
Chemotherapy (Surgical and medical procedures) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib + mFOLFOX6 (N=177) | Bevacizumab + mFOLFOX6 (N=87)
Diarrhoea (Gastrointestinal disorders) | 101 | 49
Nausea (Gastrointestinal disorders) | 97 | 47
Vomiting (Gastrointestinal disorders) | 59 | 24
Constipation (Gastrointestinal disorders) | 50 | 32
Abdominal pain (Gastrointestinal disorders) | 42 | 16
Stomatitis (Gastrointestinal disorders) | 36 | 14
Dyspepsia (Gastrointestinal disorders) | 23 | 9
Abdominal pain upper (Gastrointestinal disorders) | 13 | 8
Aphthous stomatitis (Gastrointestinal disorders) | 9 | 1
Dry mouth (Gastrointestinal disorders) | 9 | 2
Dysphagia (Gastrointestinal disorders) | 9 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 5
Flatulence (Gastrointestinal disorders) | 6 | 5
Fatigue (General disorders) | 95 | 45
Mucosal inflammation (General disorders) | 40 | 28
Asthenia (General disorders) | 37 | 17
Pyrexia (General disorders) | 17 | 13
Oedema peripheral (General disorders) | 14 | 6
Temperature intolerance (General disorders) | 11 | 9
Infusion related reaction (General disorders) | 9 | 3
Pain (General disorders) | 5 | 5
Chest pain (General disorders) | 2 | 5
Neuropathy peripheral (Nervous system disorders) | 74 | 34
Paraesthesia (Nervous system disorders) | 46 | 20
Headache (Nervous system disorders) | 28 | 12
Dysgeusia (Nervous system disorders) | 26 | 18
Peripheral sensory neuropathy (Nervous system disorders) | 21 | 13
Dizziness (Nervous system disorders) | 17 | 6
Dysaesthesia (Nervous system disorders) | 12 | 5
Lethargy (Nervous system disorders) | 11 | 3
Neurotoxicity (Nervous system disorders) | 10 | 3
Hypoaesthesia (Nervous system disorders) | 5 | 5
Amnesia (Nervous system disorders) | 1 | 5
Neutropenia (Blood and lymphatic system disorders) | 93 | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 54 | 13
Anaemia (Blood and lymphatic system disorders) | 20 | 9
Leukopenia (Blood and lymphatic system disorders) | 19 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 42 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Decreased appetite (Metabolism and nutrition disorders) | 63 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 2
Dehydration (Metabolism and nutrition disorders) | 10 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 5
Hypertension (Vascular disorders) | 77 | 25
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 34 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 14
Rash (Skin and subcutaneous tissue disorders) | 16 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 5
Urinary tract infection (Infections and infestations) | 19 | 11
Nasopharyngitis (Infections and infestations) | 8 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Weight decreased (Investigations) | 34 | 7
Neutrophil count decreased (Investigations) | 14 | 8
Alanine aminotransferase increased (Investigations) | 10 | 3
Aspartate aminotransferase increased (Investigations) | 10 | 4
Platelet count decreased (Investigations) | 10 | 3
Blood thyroid stimulating hormone increased (Investigations) | 9 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Insomnia (Psychiatric disorders) | 23 | 15
Anxiety (Psychiatric disorders) | 8 | 6
Proteinuria (Renal and urinary disorders) | 19 | 5
Hypothyroidism (Endocrine disorders) | 25 | 1
Conjunctivitis (Eye disorders) | 3 | 5
Hypersensitivity (Immune system disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or after 18 months after database lock, whichever comes first. Sponsor must receive a site's manuscript at least 30 days prior to publication for review and comment. Sponsor may delay the publication for up to 60 days to seek patent protection.